CLINICAL TRIAL: NCT05411458
Title: Effects of Telerehabilitation Programs Including Aerobic Exercise and Relaxation Training in Patients With Type-2 Diabetes With and Without COVID-19
Brief Title: Effects of Telerehabilitative Aerobic and Relaxation Exercises Patients With Type 2 Diabetes With and Without COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IzmirBozyaka-HayriyeYILMAZ-002
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Type 2 Diabetes Mellitus
Keywords: COVID-19; Type 2 Diabetes Mellitus; relaxation exercises; aerobic exercise; Hb A1c; Anxiety; Stress
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2; Anxiety Disorders

STUDY DESIGN:
Masking Description: An experimental study with a randomized controlled crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group consists of 15 Type-2 DM patients who applied for routine outpatient follow-up in the internal medicine clinic, whose diabetes tests and treatments were arranged by an internist, who had COVID-19 at least 3 months ago.
  12-week treatment program; A - 6 weeks of aerobic exercise (AE) (outdoor walking program) 6 week program B - Jacobson Progressive Relaxation Exercises (JIGE) (done by patients at home). The 6-week B program (JIGE) was applied in addition to the aerobic exercise (AE) program.
  An exercise program is 30-45 minutes, and the applications are done every other day and 3 days a week.The treatment programs started with the evaluation of the cases by the physiotherapist and are followed up using the Telerehabilitation method. At the beginning of each week, the patients were called and checked, and their exercise treatments were completed at the end of 12 weeks.
  Interventions: Other: Aerobic and Relaxation Exercises
- Control Group (Other): Control group consists of 15 Type-2 DM patients without COVID-19, who applied to the internal medicine outpatient clinic for routine outpatient follow-up, whose diabetes examinations and treatments were arranged by an internist.
  12-week treatment program; A - 6 weeks of aerobic exercise (AE) (outdoor walking program) 6 week program B - Jacobson Progressive Relaxation Exercises (JIGE) (done by patients at home). The 6-week B program (JIGE) was applied in addition to the aerobic exercise (AE) program.
  An exercise program is 30-45 minutes, and the applications are done every other day and 3 days a week.The treatment programs started with the evaluation of the cases by the physiotherapist and are followed up using the Telerehabilitation method. At the beginning of each week, the patients were called and checked, and their exercise treatments were completed at the end of 12 weeks.
  Interventions: Other: Aerobic and Relaxation Exercises

INTERVENTIONS:
Other: Aerobic and Relaxation Exercises — 12-week treatment program; A - 6 weeks of aerobic exercise (AE) (outdoor walking program) 6 week program B - Jacobson Progressive Relaxation Exercises (JIGE) (done by patients at home). The 6-week B program (JIGE) was applied in addition to the aerobic exercise (AE) program.
  Aerobic exercise (AE) program:The aerobic training program was applied as walking for 40 minutes in the open air. The Rating of Perceived Exertion (RPE) Borg Scale (6-20) was used to determine the walking pace, and they were asked to walk according to the light (11-12) level according to the Borg scale.
  An exercise program is 30-45 minutes, and the applications are done every other day and 3 days a week.The treatment programs started with the evaluation of the cases by the physiotherapist and are followed up using the Telerehabilitation method. At the beginning of each week, the patients were called and checked, and their exercise treatments were completed at the end of 12 weeks.

SUMMARY:
Type-2 Diabetes Mellitus (DM) disease, like other chronic diseases, is a group of diseases that are adversely affected by the COVID-19 pandemic.This study was planned to examine the effect of COVID-19 disease on patients with Type-2 DM and to investigate the effects of progressive relaxation exercises to be given as tele-rehabilitative on stress, anxiety and blood glucose levels and HbA1c value.

DETAILED DESCRIPTION:
30 Type-2 DM patients whose diabetes examinations and treatments were performed by an internist in the internal medicine outpatient clinic of Izmir Bozyaka Training and Research Hospital will be included in the study. (study group: 15 cases who had COVID-19 at least three months ago and control group: 15 cases who did not have COVID-19) Physical characteristics such as age (year), gender, body weight (kg), height (cm), body mass index (kg/m2) and sociodemographic characteristics of the cases were questioned. Evaluated by anthropometric measurements (waist and hip circumference (cm) and waist and body composition measurement (Xiaomi MI scale 2).

Diabetes knowledge levels were determined by the Diabetes Knowledge Test (DKT2), physical activity levels were determined by the International Physical Activity Questionnaire-Short form (IPAQ-short form), and sleep quality was determined by the Pittsburg Sleep Quality Index (PUKI). Blood values such as fasting blood glucose (mg/dl), Glycosylated Hemoglobin (HbA1c) (%) of the cases were measured, and the patient was taught to measure the heart rate (beats/minute) in a radial way. Functional capacity levels were determined by the 6-minute walking test (6MWT), lower extremity muscle strength by the Five-Time Sitting Stand Up Test (FTSST), stress levels by the Perceived Stress Scale (PSS) and anxiety levels by Spielberg's State-Trait Anxiety Inventory (STAI-S and T). ) were evaluated with Quality of life was measured with the Short Form-12 (SF-12) and Diabetes-Specific Quality of Life Scale (DQOL).

All evaluations were made face to face with all cases in both groups at the beginning of the study. Then, the same exercise training was applied to the patients in both groups as rehabilitative, in a crossover design, in a random order determined by the lottery for a total of 12 weeks.

12-week treatment program A - 6 weeks of Aerobic exercise (AE) (outdoor walking program) B - 6 week program - Jacobson Progressive Relaxation Exercises (JIGE) (performed by patients at home) were administered in addition to aerobic exercise (AE) (outdoor walking program).

The exercise program is 30-45 minutes and the applications are done every other day and 3 days a week. Patients recorded their Heart Rate (beats/minute) before and after each administration.

The Five Times Standing Test (FTSST) and STAI-S were performed at 6 weeks following treatment (at treatment changes). At the end of the treatment, that is, at the 12th week; 6 DYT and Five Time Sit to Stand Test (FTSST) and IPAQ-short form, SF-12 and DQOL, PSS, STAI-S and T, PUKI scales were re-evaluated. The efficacy of treatments will be compared within and between groups using appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

1.Volunteer patients diagnosed with Type-2 DM by a specialist 2.18 to 65 years of age 3.To have control of comorbid diseases in the last 3 months 4.Not having any condition that prevents exercise 5.Voluntarily exercising three days a week

Study group cases (for cases who have had Covid-19 Disease) in addition to the above-mentioned criteria;

1. Having had COVID-19 at least 1 time in the last 3 months
2. Having had COVID-19 at least 1 time in the last 3 months and survived the symptoms of the disease without mechanical ventilator support -

Exclusion Criteria:

1. Having additional complications such as diabetic neuropathy, nephropathy, and retinopathy
2. Having a health problem (orthopedic, neurological, internal and cardiorespiratory) that prevents standing up / walking
3. no internet connection
4. malignancy, acute inflammation, intestinal tumor
5. Having cognitive impairment, vision and hearing loss that may interfere with working -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from Baseline in HbA1c at 12 weeks
  HbA1c test, also known as the haemoglobin A1c or glycated haemoglobin test, is an important blood test that gives a good indication of how well your diabetes is being controlled
Fasting blood sugar | Change from Baseline in fasting blood sugar at 12 weeks
  Expected values as a result of fasting blood glucose measurement range from 70 mg/dL (3.9 mmol/L) to 100 mg/dL (5.6 mmol/L).
Exercise capacity | Change from Baseline in 6 DMW at 12 weeks
  The 6-min walk (6MW) test is commonly used to assess exercise capacity in patients and to track functional change resulting from disease progression or therapeutic intervention.
anxiety | Change from Baseline in STAI-S and T at 6 and 12 weeks
  Spielberg State-Trait Anxiety Inventory (STAI-S and T) was used to assess anxiety. The total score obtained from the scale varies between 20-80. A high score indicates a high level of anxiety.
Lower limb Strength | Change from Baseline in FTSST at 6 and 12 weeks
  The Five Time Sit to Stand Test (FTSST) is used to measure a patient's functional mobility and muscle strength of their lower extremities.
Physical Activity | Change from Baseline in IPAQ at 12 weeks
  The International Physical Activity Questionnaire (IPAQ) is a frequently used instrument for the evaluation of physical activity (PA). It was developed in order to assess physical activity in adults aged 18-65 years
Stress | Change from Baseline in PSS at 12 weeks
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful.
Heart rates | Change from Baseline in heart rates at 12 weeks
  Heart rates(beats/min) were measured before and after treatments. Measurements were made by the method of measuring the individual's own heart rate from the radial artery. Normal resting heart rate for adults ranges from 60 to 100 beats per minute.

SECONDARY OUTCOMES:
Sleep quality | Change from Baseline in PSQI at 12 weeks
  Petersburg sleep quality index (PSQI), PSQI is a eighteen item scale.The total scores range is 0-21. A higher score indicates a worse sleep quality.
Health Related Quality of Life | Change from Baseline in SF-12 at 12 weeks
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet G KARAKAYA, Prof, PT, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Hayriye Yılmaz, Izmir, Turkey (Türkiye)